CLINICAL TRIAL: NCT04215601
Title: Effect of Phototherapy on Serum Level of Calcium in Infants With Hyperbilirubinemia
Brief Title: Effect of Phototherapy on Serum Calcium
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, A.L.Mohamed, Resident doctor, Assiut University
Other Study IDs: pt effect on calcium
Record Dates: First submitted 2019-12-29; First posted 2020-01-02 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Phototherapy; Side Effects
Keywords: phototherapy; hypocalcemia
MeSH Terms: conditions — Hypocalcemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Days
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Through this study our aim was to evaluate whether significant change in serum calcium level occurs in term newborns who are undergoing phototherapy and to find out the association between effect of phototherapy on serum calcium level and birth weight, postnatal age and type of feeding.

DETAILED DESCRIPTION:
Jaundice is the yellow discoloration of skin, sclerae, and other tissues caused by the deposition of bilirubin.

Approximately 60% of term and 80% of preterm babies develop jaundice in the first week of life, and about 10% of breastfed babies are still jaundiced at 1 month. Jaundice is a common cause of readmission to hospital after early discharge of newborn infants.

The most common form of hyperbilirubinaemia observed in neonates is due to unconjugated or unbound bilirubin. High levels of unconjugated bilirubin are managed by treatment of the underlying cause (e.g. dehydration and sepsis), provision of phototherapy, administration of immunoglobulin (in certain cases of haemolytic anaemia) and, in very severe cases, exchange transfusion. If left untreated, extreme elevation of unconjugated bilirubin can lead to permanent brain damage (kernicterus) and/or death.

However, exchange transfusion is associated with a significant morbidity, and even mortality while phototherapy has several disadvantages which include increasing the duration of hospitalization, costs and mother-child separation . It also has some reported side effects as rash, loose green stools, dehydration, ocular hazards, oxidative injury, hyperthermia and water loss and may be associated with some long-term side effects such as melanocytic nevi, skin cancer, allergic disease, patent ductus arterious and retinal damage .

Some studies are available concerning the prevalence of hypocalcemia in neonates after phototherapy, but the results varied based on where the studies were conducted. So, more studies were required to reach a definite conclusion. Through this study our aim was to evaluate whether significant change in serum calcium level occurs in term newborns who are undergoing phototherapy and to find out the association between effect of phototherapy on serum calcium level and birth weight, postnatal age and type of feeding.

ELIGIBILITY:
Inclusion Criteria:

* Stable term neonates with jaundice who require management with phototherapy and are fed with full strength formula or breast fed.

Exclusion Criteria:

* Jaundiced neonates with hypocalcemia.
* Jaundiced neonates needing exchange transfusion.
* Jaundiced neonates suffering from hypothyroidism.
* Jaundiced infants of diabetic mother.
* Jaundiced infants with other illness as severe RDS, perinatal asphyxia,Sever sepsis or hemolytic disease of newborn.
* Jaundiced infants with congenital abnormalities.

Ages: 1 Hour to 30 Days | Sex: All
Age Groups: Child
Study Population: Infants who will come at neonatal unit of Assiut University Children's Hospital meeting our inclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2022-02-10 (Actual); Study Completion 2022-02-20 (Actual)

PRIMARY OUTCOMES:
Serum calcium level after 48 hours of phototherapy | 2days
  The neonates under study will be compared regarding serum bilirubin level and serum calcium level prior to start of study and then repeated after 48 hours to show any significant change in serum calcium level after exposure to phototherapy

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut children's hospital, Asyut, Egypt

REFERENCES:
- [Background] Amos RC, Jacob H, Leith W. Jaundice in newborn babies under 28 days: NICE guideline 2016 (CG98). Arch Dis Child Educ Pract Ed. 2017 Aug;102(4):207-209. doi: 10.1136/archdischild-2016-311556. Epub 2017 Feb 8. No abstract available. PMID 28179382
- [Background] Alizadeh-Taheri P, Sajjadian N, Eivazzadeh B. Prevalence of phototherapy induced hypocalcemia in term neonate. Iran J Pediatr. 2013 Dec;23(6):710-1. No abstract available. PMID 24910756
- [Background] Shahriarpanah S, Haji Ebrahim Tehrani F, Davati A, Ansari I. Effect of Phototherapy on Serum Level of Calcium, Magnesium and Vitamin D in Infants With Hyperbilirubinemia. Iran J Pathol. 2018 Summer;13(3):357-362. Epub 2018 Sep 12. PMID 30636959
- [Background] Hansen TW. [Treatment of neonatal jaundice]. Tidsskr Nor Laegeforen. 2005 Mar 3;125(5):594-8. Norwegian. PMID 15776035
- [Background] Waterham M, Bhatia R, Donath S, Molesworth C, Tan K, Stewart M. Phototherapy in transport for neonates with unconjugated hyperbilirubinaemia. J Paediatr Child Health. 2016 Jan;52(1):67-71. doi: 10.1111/jpc.12984. Epub 2015 Aug 19. PMID 26289553
- [Background] Xiong T, Tang J, Mu DZ. [Side effects of phototherapy for neonatal hyperbilirubinemia]. Zhongguo Dang Dai Er Ke Za Zhi. 2012 May;14(5):396-400. Chinese. PMID 22613117
- [Background] Kargar M, Jamshidi Z, Beheshtipour N, Pishva N, Jamali M. Effect of head covering on phototherapy-induced hypocalcaemia in icterus newborns; a randomized controlled trial. Int J Community Based Nurs Midwifery. 2014 Apr;2(2):121-6. PMID 25349853